CLINICAL TRIAL: NCT04675879
Title: Clinical and Radiological Results of Conservative Treatments in Proximal Humerus Fractures.Prospective Randomized Trial
Brief Title: Clinical and Radiological Results of Conservative Treatments in Proximal Humerus Fractures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Murat Sarikas, Recident of orthopaedic surgery, Bezmialem Vakif University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 14052
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Proximal Humeral Fracture
Keywords: proximal humeral fractures; conservative treatments
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Intervention Model Description: Previously randomized patients were divided into 3 groups to be treated with 3 different types of bandages.
Who Masked: Investigator, Outcomes Assessor
Masking Description: When the treatments are completed, those who will evaluate the clinical and radiological results will not know the treatment method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Velpau bandage (Group 1) (Experimental): Patients with neer type 2, 3 or 4 proximal humerus fractures under conservative follow-up with velpau bandage.
  Interventions: Device: Shoulder arm bandage
- Shoulder arm sling (Group 2) (Experimental): Patients with neer type 2, 3 or 4 proximal humerus fractures under conservative follow-up with shoulder arm sling.
  Interventions: Device: Shoulder arm bandage
- Padded shoulder arm sling (Group 3) (Experimental): Patients with neer type 2, 3 or 4 proximal humerus fractures under conservative follow-up with padded shoulder arm sling with 30 degree abduction.
  Interventions: Device: Shoulder arm bandage

INTERVENTIONS:
Device: Shoulder arm bandage — Three different shoulder-arm bandage types

SUMMARY:
In the investigators' prospective randomized study, the investigator will investigate the effect of different bandage types on functional and radiological results of proximal humerus fractures over 18 years of age, for whom conservative treatment is decided.

In recent studies, it has been shown that surgical treatment in proximal humerus fractures has a high complication rate and is also not superior to conservative treatments in terms of functional results. Therefore, the importance of conservative treatment is increasing day by day in this group of fractures, especially in elderly patients with high risk for surgery.

In these studies in the literature, the method in conservative treatment is not clearly specified, and the investigator will apply 3 different bandages to adjust the rotation of the shoulder in 3 different ways during the investigators' conservative treatment. The investigator will compare functional and radiological results between these groups.

DETAILED DESCRIPTION:
Proximal humerus fractures, who are admitted to the investigators' emergency department and are decided to follow conservative follow-up criteria, will be given one of 3 different bandages (velpau bandage, classical shoulder arm sling, 30 degree padded shoulder arm sling) according to the previous randomization.

Routinely, at the 2nd week, 6th week, 12th week, 6th month and 12th month outpatient clinic controls, the patients will be seen and their X-ray and clinical satisfaction status will be checked. X-rays will be taken as classical ap / lateral and true ap.

At the end of the second week, which is absolute immobilization, elbow and wrist movements will begin. Afterwards, in the 6th week, according to the state of union with deltoid strengthening, passive and active shoulder joint range of motion exercises will be started.

At the end of the 12th month, the follow-up will be terminated, and in this control, the existing joint movements will be recorded by measuring the degrees of anterior elevation, abduction, external rotation in neutral, external rotation at 90 degrees and internal rotation. In addition, in this control, the values will be noted by taking the Constant, ASES, DASH and VAS Scores.

After all these values are noted for all 3 groups, statistical analysis between groups will be made for each variable and the result will be given.

In addition, if complications(non-union,mal-union,stiffness etc.) occur during conservative follow-up in the investigators' patients, they will be recorded and whether there is a statistically significant difference in complications between the groups will be investigated.

The investigators' aim in this study is to understand whether any of these 3 different bandage types, which are routinely used as an immobilization method in proximal humerus fractures, are superior to the other.

A study comparing immobilization methods could not be found in the literature. These bandage types, which have not been compared with their effectiveness, are used effectively all over the world. With this study, the investigator set this on a scientific basis and set the correct direction of the investigators' treatments as the investigators' main goal.

ELIGIBILITY:
Inclusion Criteria:

* Neer type 2, 3 and 4 proximal humerus fractures suitable for conservative follow-up
* Patients older than 18 years

Exclusion Criteria:

* Previous surgery in the ipsilateral shoulder area
* Fractured dislocation
* Patients with open phys line
* Patients with neurological problems affecting the upper extremity (MS, stroke, etc.)
* Patients with fracture-induced neurovascular problems
* Open fractures
* Patients who require surgery for any reason while follw-up (malunion, nonunion, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
External rotation degree | 12 months
  degrees of external rotation achieved after conservative follow-up.

SECONDARY OUTCOMES:
Anterior elevation degree | 12 months
  degrees of anterior elevation achieved after conservative follow-up.
Abduction degree | 12 months
  degrees of abduction achieved after conservative follow-up.
Internal rotation degree | 12 months
  degrees of internal rotation achieved after conservative follow-up.
DASH Score degree | 12 months
  DASH score obtained at the end of follow-up of patients who completed 12 months of conservative follow-up.
  Minimum and maximum values are respectively 0 and 100. Higher scores mean a worse outcome.
Constant Score degree | 12 months
  Constant score obtained at the end of follow-up of patients who completed 12 months of conservative follow-up Minimum and maximum values are respectively 8 and 100. Higher scores mean a better outcome.
ASES Score degree | 12 months
  ASES score obtained at the end of follow-up of patients who completed 12 months of conservative follow-up Minimum and maximum values are respectively 0 and 100. Higher scores mean a better outcome.
VAS Score degree | 12 months
  VAS score obtained at the end of follow-up of patients who completed 12 months of conservative follow-up Minimum and maximum values are respectively 0 and 10. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kapıcıoğlu, Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
How many patients have been followed up so far?
Supporting Information: CSR
Time Frame: 3 months
Access Criteria: 6 months and 9 months after the start of the study. June 8 : The number of patients with follow-up reached 45. The 3rd month examinations were performed on half of our patients.

REFERENCES:
- See also: Manuel Soler-Peiro , Lorena García-Martínez , Luis Aguilella and Marcelino Perez-Bermejo . Conservative treatment of 3-part and 4-part proximal humeral fractures: a systematic review . Soler-Peiro et al. Journal of Orthopaedic Surgery and Research — https://doi.org/10.1186/s13018-020-01880-7
- See also: Operative versus non-operative treatment for 2-part proximal humerus fracture: A multicenter randomized controlled trial . PLOS Medicine — https://doi.org/10.1371/journal.pmed.1002855
- See also: Lisa Howard , Randa Berdusco , Franco Momoli , J. Pollock , Allan Liew , Steve Papp , Karl-Andre Lalonde , Wade Gofton , Sara Ruggiero and Peter Lapner . Open reduction internal fixation vs non- operative management in proximal humerus fractures: a prosp — https://doi.org/10.1186/s12891-018-2223-3